CLINICAL TRIAL: NCT00556608
Title: Efficacy Evaluation of Intra-articular Hyaluronic Acid (Sinovial®) vs Synvisc® in the Treatment of Symptomatic Knee Osteoarthritis. A Double-blind, Controlled, Randomised, Parallel-group Non-inferiority Study
Brief Title: Efficacy Study of Intra-articular Hyaluronic Acid in the Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06CZIFCH/Hai06
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sinovial (Experimental): 3 intra-articular injections of Sinovial®
  Interventions: Device: Sinovial® (syringe containing sodium hyaluronate solution)
- Sinvisc (Active Comparator)
  Interventions: Device: Synvisc® ( syringe containing Hylan G-F 20 solution)

INTERVENTIONS:
Device: Sinovial® (syringe containing sodium hyaluronate solution) — 2 mL 0.8% sodium hyaluronate (16 mg) solution. 3 intra-articular injections once-a-week.
  Other Names: Sinovial®: Class III medical device(CE mark n° 0499)
  Arms: Sinovial
Device: Synvisc® ( syringe containing Hylan G-F 20 solution) — 2 mL 0.8% Hylan G-F 20 (16 mg) solution. 3 intra-articular injections once-a-week.
  Other Names: Synvisc®: class III medical device (CE mark n° 0088)
  Arms: Sinvisc

SUMMARY:
The purpose of this study is to prove the non-inferiority of the intra-articular injection of hyaluronic acid (Sinovial®) in the symptomatic treatment of knee OA in comparison to Synvisc®.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years
* Primary knee OA of the medial or lateral femoro-tibial compartment
* Symptoms for at least 3 months
* Diagnosis according to ACR criteria
* Kellgren & Lawrence radiological grade 2-3
* Patients who failed to respond sufficiently (not responders) to analgesics and/or NSAIDs taken regularly or responders intolerant to the regular use of analgesics and/or NSAIDs.
* Mean WOMAC pain subscore at the target knee >= 40 mm and < 80 mm on a VAS at baseline after wash-out from analgesics/NSAIDs· If bilateral knee OA: definition of the most symptomatic joint at screening based on patient's evaluation and Investigator's clinical judgment and mean WOMAC pain subscore at baseline in the contra-lateral knee < 30 mm
* Written informed consent
* Subject able to understand, co-operative and reliable

Exclusion Criteria:

* BMI >= 32 kg/m2
* Secondary (post-traumatic) knee OA
* Predominantly patello-femoral pain/syndrome
* No remaining joint space width
* Symptomatic hip OA or other interfering health condition
* Severe varus/valgus deformity (>15°)
* History/present evidence of (target knee): inflammatory, infective or metabolic joint diseases; recurrent clinical chondrocalcinosis; crystal arthropaties; osteo-articular pathologies differing from arthrosis; articular fracture; ochronosis; acromegaly; haemochromatosis; Wilson's disease; primary osteochondromatosis; heritable disorders; collagen gene mutations.
* Concomitant rheumatic disease
* Significant injury to the target knee in the last 6 months
* Previous joint replacement/arthroplasty (target knee)
* Arthroscopy/osteotomy/surgery in the past 1 year (target knee)
* Any surgery scheduled in the next 6 months
* Venous or lymphatic stasis in the relevant limb
* Skin infection/disease/trauma at the injection site
* Systemic or i.a. (target knee) corticosteroids in the past 3 months
* I.a. corticosteroids (non-target joint) in the past 4 weeks
* Viscosupplementation (target knee) in the past year
* Recently started (in the last 3 months) physical therapy (target knee)
* Recently (in the last 3 months) started therapy or change in dosage of SYSADOAs
* Ongoing anticoagulant therapy
* Chronic or recurrent use of NSAIDs/analgesics/narcotics because of diseases different from OA of the target knee
* History of allergy or hypersensitivity to hyaluronic acid or paracetamol or avian proteins
* Participation in a clinical study in the last 3 months
* Pregnant or lactating women, and women of childbearing potential not willing to use adequate contraception
* Patients unable to stay in the study for 6 months, non-cooperating, not able to understand

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Improvement in WOMAC pain subscore from baseline | to week 26

SECONDARY OUTCOMES:
Change in WOMAC OA Index total score and pain, function and stiffness subscores;Change in Lequesne's algofunctional index; Change in global pain (visit assessment); Change in global status by the patient;Change in global status by the Investigator;SPID% | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karel PAVELKA, MD, Principal Investigator — Institute of Rheumatology-Na Slupi 4 - 12850 Praha 2 (Czech Republic)
Locations (20):
- Czechia (4):
  - Interni hemato-onkologická klinika, Fakultní nemocnice, Brno-Bohunice
  - ARTHROMED s.r.o., Pardubice
  - Institute of Rheumatology, Prague
  - Centrum léčby pohybového aparátu spol. s.r.o., Prague
- France (2):
  - University Hospital Centre Bois-Guillaume, Bois-Guillaume
  - University Hospital Centre of Limoges - Rheumatology Service, Limoges
- Germany (3):
  - Orthopädische Universitätsklinik und Poliklinik der RWTH Aachen, Aachen
  - Nova clinic, Biberach an der Riss
  - Orthopädische Praxis, Stockach
- Italy (6):
  - Sezione Dipartimentale a valenza provinciale di Reumatologia - AzUSL 8, Arezzo
  - Ospedale Privato Accreditato Nigrisoli, Bologna
  - Medicina e Traumatologia dello Sport - AzUSL 2 Lucca, Lucca
  - Unità Operativa di Reumatologia - Istituto Ortopedico Gaetano Pini, Milan
  - Rheumatology Unit Santa Chiara Hospital, Pisa
  - Unità Operativa di Reumatologia - Az. Ospedaliera Universitaria Senese - Policlinico "Le Scotte", Siena
- Slovakia (4):
  - F.D. Roosevelt's University Hospital, Banská Bystrica
  - Romjan s.r.o., Bratislava
  - National Institute of Rheumatic Diseases, Piešťany
  - Rheumatology Clinic, Reumaglobal s.r.o, Trnava
- Department of Rheumatology and Institute of Physical Medicine - Zurich University, Zurich, Switzerland

REFERENCES:
- [Background] Theiler R, Bruhlmann P. Overall tolerability and analgesic activity of intra-articular sodium hyaluronate in the treatment of knee osteoarthritis. Curr Med Res Opin. 2005 Nov;21(11):1727-33. doi: 10.1185/030079905X65547. PMID 16307692
- [Background] Castellacci E, Polieri T. Antalgic effect and clinical tolerability of hyaluronic acid in patients with degenerative diseases of knee cartilage: an outpatient treatment survey. Drugs Exp Clin Res. 2004;30(2):67-73. PMID 15272644
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000 Sep;43(9):1905-15. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-P. No abstract available. PMID 11014340
- [Background] Altman RD. Status of hyaluronan supplementation therapy in osteoarthritis. Curr Rheumatol Rep. 2003 Feb;5(1):7-14. doi: 10.1007/s11926-003-0077-6. PMID 12590879
- [Background] Lo GH, LaValley M, McAlindon T, Felson DT. Intra-articular hyaluronic acid in treatment of knee osteoarthritis: a meta-analysis. JAMA. 2003 Dec 17;290(23):3115-21. doi: 10.1001/jama.290.23.3115. PMID 14679274
- [Background] Wang CT, Lin J, Chang CJ, Lin YT, Hou SM. Therapeutic effects of hyaluronic acid on osteoarthritis of the knee. A meta-analysis of randomized controlled trials. J Bone Joint Surg Am. 2004 Mar;86(3):538-45. doi: 10.2106/00004623-200403000-00012. PMID 14996880
- [Background] Bellamy N, Campbell J, Robinson V, Gee T, Bourne R, Wells G. Viscosupplementation for the treatment of osteoarthritis of the knee. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD005321. doi: 10.1002/14651858.CD005321.pub2. PMID 16625635
- [Background] Recommendations for the registration of drugs used in the treatment of osteoarthritis. Group for the respect of ethics and excellence in science (GREES): osteoarthritis section. Ann Rheum Dis. 1996 Aug;55(8):552-7. doi: 10.1136/ard.55.8.552. No abstract available. PMID 8774185
- [Background] Altman R, Brandt K, Hochberg M, Moskowitz R, Bellamy N, Bloch DA, Buckwalter J, Dougados M, Ehrlich G, Lequesne M, Lohmander S, Murphy WA Jr, Rosario-Jansen T, Schwartz B, Trippel S. Design and conduct of clinical trials in patients with osteoarthritis: recommendations from a task force of the Osteoarthritis Research Society. Results from a workshop. Osteoarthritis Cartilage. 1996 Dec;4(4):217-43. doi: 10.1016/s1063-4584(05)80101-3. No abstract available. PMID 11048620
- [Background] Strand V, Kelman A. Outcome measures in osteoarthritis: randomized controlled trials. Curr Rheumatol Rep. 2004 Feb;6(1):20-30. doi: 10.1007/s11926-004-0080-6. PMID 14713399
- [Background] Kirchner M, Marshall D. A double-blind randomized controlled trial comparing alternate forms of high molecular weight hyaluronan for the treatment of osteoarthritis of the knee. Osteoarthritis Cartilage. 2006 Feb;14(2):154-62. doi: 10.1016/j.joca.2005.09.003. Epub 2005 Oct 19. PMID 16242361
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Bellamy N. WOMAC: a 20-year experiential review of a patient-centered self-reported health status questionnaire. J Rheumatol. 2002 Dec;29(12):2473-6. No abstract available. PMID 12465137
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Lockman LE. Practice tips. Knee joint injections and aspirations: the triangle technique. Can Fam Physician. 2006 Nov;52(11):1403-4. No abstract available. PMID 17279197
- [Background] Lequesne MG, Mery C, Samson M, Gerard P. Indexes of severity for osteoarthritis of the hip and knee. Validation--value in comparison with other assessment tests. Scand J Rheumatol Suppl. 1987;65:85-9. doi: 10.3109/03009748709102182. PMID 3479839
- [Background] Lequesne M, Samson M, Gerard P, Mery C. [Pain-function indices for the follow-up of osteoarthritis of the hip and the knee]. Rev Rhum Mal Osteoartic. 1990 Oct 30;57(9 ( Pt 2)):32S-36S. French. PMID 2080414
- [Background] Ali Y, Weinstein M, Jokl P. Acute pseudogout following intra-articular injection of high molecular weight hyaluronic acid. Am J Med. 1999 Dec;107(6):641-2. doi: 10.1016/s0002-9343(99)00255-7. No abstract available. PMID 10625037
- [Background] Luzar MJ, Altawil B. Pseudogout following intraarticular injection of sodium hyaluronate. Arthritis Rheum. 1998 May;41(5):939-40. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-D. No abstract available. PMID 9588748
- [Background] Maillefert JF, Hirschhorn P, Pascaud F, Piroth C, Tavernier C. Acute attack of chondrocalcinosis after an intraarticular injection of hyaluronan. Rev Rhum Engl Ed. 1997 Oct;64(10):593-4. No abstract available. PMID 9385702
- [Background] Allen E, Krohn K. Adverse reaction to Hylan GF-20. J Rheumatol. 2000 Jun;27(6):1572. No abstract available. PMID 10852302
- [Background] Chen AL, Desai P, Adler EM, Di Cesare PE. Granulomatous inflammation after Hylan G-F 20 viscosupplementation of the knee : a report of six cases. J Bone Joint Surg Am. 2002 Jul;84(7):1142-7. PMID 12107313
- [Background] Zardawi IM, Chan I. Synvisc perisynovitis. Pathology. 2001 Nov;33(4):519-20. doi: 10.1080/00313020120083296. PMID 11827424
- [Background] Hamburger MI, Lakhanpal S, Mooar PA, Oster D. Intra-articular hyaluronans: a review of product-specific safety profiles. Semin Arthritis Rheum. 2003 Apr;32(5):296-309. doi: 10.1053/sarh.2002.50008. PMID 12701040
- [Background] Ehrich EW, Davies GM, Watson DJ, Bolognese JA, Seidenberg BC, Bellamy N. Minimal perceptible clinical improvement with the Western Ontario and McMaster Universities osteoarthritis index questionnaire and global assessments in patients with osteoarthritis. J Rheumatol. 2000 Nov;27(11):2635-41. PMID 11093446
- [Background] Angst F, Aeschlimann A, Michel BA, Stucki G. Minimal clinically important rehabilitation effects in patients with osteoarthritis of the lower extremities. J Rheumatol. 2002 Jan;29(1):131-8. PMID 11824949
- [Background] Bijlsma JW. Patient centred outcomes in osteoarthritis. Ann Rheum Dis. 2005 Jan;64(1):1-2. doi: 10.1136/ard.2004.025072. No abstract available. PMID 15608297
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Derived] Pavelka K, Uebelhart D. Efficacy evaluation of highly purified intra-articular hyaluronic acid (Sinovial((R))) vs hylan G-F20 (Synvisc((R))) in the treatment of symptomatic knee osteoarthritis. A double-blind, controlled, randomized, parallel-group non-inferiority study. Osteoarthritis Cartilage. 2011 Nov;19(11):1294-300. doi: 10.1016/j.joca.2011.07.016. Epub 2011 Aug 16. PMID 21875678